CLINICAL TRIAL: NCT04787913
Title: An Evaluation of a Dynamic Web-Based Visualization of Community Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: herdimm
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Vaccine-Preventable Diseases
Keywords: herd immunity; community immunity; web-based application; visualization
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Intervention Model Description: This study will be a multi-armed factorial randomized controlled trial. Each participant will be randomly allocated to focus on one of four possible vaccine-preventable diseases: measles, pertussis, flu (influenza), or a generic vaccine-preventable disease (hereby referred to as "generic"). All aspects of the study (visualization, questionnaire) will be focused on that one disease for that participant. The primary and secondary outcomes of the study which are risk perception, emotion, knowledge, trust in information provided, attitudes and a validated scale about vaccination (Betsch et al. 2018) will be assessed in an online questionnaire.
  Because three online visualizations are available only in English whereas our study will be conducted in both English and French, we will use slightly different randomization patterns for English- and French-speaking participants.
Who Masked: Investigator
Masking Description: This will be a single-blinded study because we cannot mask participants to the fact that they have been randomized to a visualization e.g., about measles. However, participants will not necessarily know the purpose of the study arm to which they are assigned,and investigators will be blinded to study arm during data analysis (investigators are not aware of whether the next eligible participant will be receiving treatment or control intervention.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- controlgeneric (No Intervention): No intervention provided. Participant answers outcome questions about an unnamed vaccine-preventable disease. English and French.
- controlmeasles (No Intervention): No intervention provided. Participant answers outcome questions about measles. English and French.
- controlpertussis (No Intervention): No intervention provided. Participant answers outcome questions about pertussis. English and French.
- controlflu (No Intervention): No intervention provided. Participant answers outcome questions about flu. English and French.
- herdimmgeneric (Experimental): Web-based application (main intervention) provided. Participant answers outcome questions about an unnamed vaccine-preventable disease. English and French.
  Interventions: Behavioral: herdimm
- herdimmmeasles (Experimental): Web-based application (main intervention) provided. Participant answers outcome questions about measles. English and French.
  Interventions: Behavioral: herdimm
- herdimmpertussis (Experimental): Web-based application (main intervention) provided. Participant answers outcome questions about pertussis. English and French.
  Interventions: Behavioral: herdimm
- herdimmflu (Experimental): Web-based application (main intervention) provided. Participant answers outcome questions about flu. English and French.
  Interventions: Behavioral: herdimm
- robertkochgeneric (Active Comparator): Web-based application (comparator) provided. Participant answers outcome questions about an unnamed vaccine-preventable disease. English only.
  Interventions: Behavioral: robertkochgeneric
- sbsnewsgeneric (Active Comparator): Video (comparator) provided. Participant answers outcome questions about an unnamed vaccine-preventable disease. English only.
  Interventions: Behavioral: sbsnewsgeneric
- guardianmeasles (Active Comparator): Video (comparator) provided. Participant answers outcome questions about measles. English only.
  Interventions: Behavioral: guardianmeasles
- theotheredmundmeasles (Active Comparator): Video (comparator) provided. Participant answers outcome questions about measles. English only.
  Interventions: Behavioral: theotheredmundmeasles
- publichealthagencycanadaflu (Active Comparator): Video (comparator) provided. Participant answers outcome questions about flu. English and French.
  Interventions: Behavioral: publichealthagencycanadaflu

INTERVENTIONS:
Behavioral: herdimm — In this visualization participants can build their own avatar representing themselves and 8 other avatars representing people around them, like their family or coworkers. Our visualization then uses these avatars in a brief narrated video explaining how herd immunity works.
  Arms: herdimmflu; herdimmgeneric; herdimmmeasles; herdimmpertussis
Behavioral: guardianmeasles — A screen capture of an interactive visualization: https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated
  Arms: guardianmeasles
Behavioral: theotheredmundmeasles — A gif showing measles spreading through populations with differing levels of vaccine coverage: https://imgur.com/gallery/8M7q8#J7LANQ4
  Arms: theotheredmundmeasles
Behavioral: sbsnewsgeneric — A video showing how herd immunity works in general: https://www.sbs.com.au/news/two-sydney-babies-too-young-to-be-vaccinated-infected-with-measles
  Arms: sbsnewsgeneric
Behavioral: publichealthagencycanadaflu — A video showing how herd immunity works in the context of influenza: https://www.canada.ca/fr/sante-publique/services/video/la-grippe-n-en-passez-pas-les-maux.html
  Arms: publichealthagencycanadaflu
Behavioral: robertkochgeneric — A web-based application showing how herd immunity works in general: http://rocs.hu-berlin.de/D3/herd/
  Arms: robertkochgeneric

SUMMARY:
This study is a PhD project conducted by Ms. Hina Hakim, supervised by Dr. Holly O. Witteman, PhD, and co-supervised Dr. Daniel Reinharz, professors and researchers at the Faculty of Medicine at Laval University. The purpose of this study is to evaluate the effects of visualization conveying the concept of community immunity or herd immunity on risk perception (towards individual, family, community and vulnerable people in communities) (primary outcome) and on emotions, attitudes, knowledge, and behavioural intentions (secondary outcomes).

DETAILED DESCRIPTION:
Visualization is a powerful communication mechanism that uses pre-attentive processing to communicate large amounts of information rapidly in understandable and compelling ways (Healey and Enns 2012). A systematic review demonstrates that there are some interventions available for conveying the concept of community immunity, and very few evaluate interventions for their effects on vaccine intentions and uptake as well as their precursors, such as knowledge, attitudes, knowledge and none on emotions (Hakim et al. 2018).

The purpose of this study is to evaluate the effects of visualization conveying the concept of community immunity on risk perception (to individual, family, community and vulnerable people in communities) (primary outcome) and on emotions, attitudes, knowledge, and behavioural intentions (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Members of the general population in Canada
* At least 18 years old
* Able to provide free and informed consent
* Able to read and understand French or English
* Able to use a computer

Exclusion Criteria:

- No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5516 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Risk perception | immediately after intervention or control
  6 items assessing risk perception (item 1 = risk perception as comprehension, scale 0-100, higher numbers better; items 2-5 = risk perception as feelings, scale 1-7, higher numbers better; complete list of items and response wording available in uploaded questionnaire herdimm_phase3_questionnaire_2021-03-01.pdf)

SECONDARY OUTCOMES:
Emotions | immediately after intervention or control
  5 items (e.g., "I am worried about getting [disease]", "I would feel guilty if a vulnerable person (a baby, a young child, an older person, a cancer patient) got [disease] from me") with a 7-point Likert-type response scale ranging from "strongly disagree" to "strongly agree"; higher numbers may be better; complete list of items and response wording available in uploaded questionnaire herdimm_phase3_questionnaire_2021-03-01.pdf
Knowledge | immediately after intervention or control
  15 items, with 2 multiple choice questions and 13 true/false questions, for a total possible score ranging from 0 to 18; higher numbers better; complete list of items available in uploaded questionnaire herdimm_phase3_questionnaire_2021-03-01.pdf
Trust in information | immediately after intervention or control
  Single item (Control: "During your life, you may have seen information about vaccines. Thinking about the information you have seen, how trustworthy was it?" Treatment: "Earlier, you saw a {{video, website}} about herd immunity. Thinking about the {{video, website}} you saw earlier, how trustworthy was the information in it?") with Likert-type response options 1 = not at all trustworthy, 2 = moderately untrustworthy, 3 = slightly untrustworthy, 4 = neutral, 5 = slightly trustworthy, 6 = moderately trustworthy, 7 = strongly trustworthy
Vaccination intentions | immediately after intervention or control
  Questions conditioned on whether the participant indicates they believe they are already immune to the disease in question, e.g., "Imagine you were not already immune to {{measles/pertussis/influenza/a vaccine preventable disease}}. If you were eligible to receive a free vaccine against {{measles/pertussis/influenza/a vaccine-preventable disease}}, how likely would you be to get vaccinated?" Response scale on a slider: 0 = extremely unlikely, I would definitely NOT be vaccinated; 100 = extremely likely, I would definitely BE vaccinated; higher numbers better.
5C scale | immediately after intervention or control
  "5C scale: 15-item validated scale measuring the psychological antecedents of vaccination (Betsch et al., 2018)"

CONTACTS AND LOCATIONS:
Overall Officials: Holly Witteman, PhD, Principal Investigator — Laval University
Locations (1):
- Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data (answers to questions in the survey including socio-demographic information) will be deposited in a public repository (Dataverse de l'Université Laval (Laval University)) which will allow data sharing with the scientific community. No information that would allow anyone to identify a person will be deposited in this public repository. Study protocol and statistical analysis plan have been deposited in Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: As soon as possible upon completion of the study and posting of a preprint with results.
Access Criteria: Freely available.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04787913/Prot_SAP_ICF_000.pdf